CLINICAL TRIAL: NCT06155448
Title: Perennial Malaria Chemoprevention (PMC) Effect Study: Nigeria Operational Feasibility and Effectiveness
Brief Title: Perennial Malaria Chemoprevention (PMC) Effect Study
Acronym: PMCEffect
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malaria Consortium (Other)
Collaborators: Nigerian Institute of Medical Research (Other Government); London School of Hygiene and Tropical Medicine (Other); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PMCEFFECTNG; INV-004302 (Other Grant/Funding Number: Bill & Melinda Gates Foundation)
Record Dates: First submitted 2023-11-14; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Malaria
Keywords: PMC; Chemoprevention; Malaria; Integrated delivery
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: The intervention arm will comprise PMC-plus: A 6-scheduled dose regimen administered to eligible children at 10 weeks, 14 weeks, 6 months, 9 months, 12 months and 15 months of age concurrently with EPI vaccinations DTP2/Penta2, DTP3/Penta3, vitamin A, and measles immunisation where appropriate. Eligible children attending the participating health facilities for other reasons beyond EPI would be invited to receive additional monthly doses between scheduled EPI-linked visits up until the child reaches 18 months of age
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PMC intervention (Experimental): The PMC intervention is designed to deliver a core regimen of six paediatric doses of sulphadoxine pyrimethamine linked to the EPI delivery platform in children 10 weeks to 15 months of age through trained health facility staff, plus additional 'pragmatic' monthly doses offered outside of the EPI schedule to children up to 18 months of age. Additional social mobilisation and social behaviour change (SBC) activities will be conducted throughout the implementation period to increase demand and uptake of vaccination and PMC services in the study population. at EPI scheduled touchpoints, plus additional monthly doses at non-scheduled monthly intervals up to age 18 months. The primary source of delivery will be government-run primary care health facilities in intervention arm wards. Coordination of implementation of the study within intervention and control arm wards will take place at the LGA level (unit of implementation).
  Interventions: Other: Perennial Malaria Chemoprevention effect
- Control (No Intervention): The control sites will have normal immunization as business as usual. However, the same sentinel site surveillance happening in the intervention arm will also be carried out in this arm. Pharmacovigilance will be passive in the control arm.

INTERVENTIONS:
Other: Perennial Malaria Chemoprevention effect — Assessing the effectiveness and feasibility of Perennial malaria chemoprevention delivery through EPI platform.
  Other Names: PMC effect
  Arms: PMC intervention

SUMMARY:
The Malaria Consortium Nigeria (MC) will coordinate a trial of PMC in Osun State, Nigeria with strategic support from the National Malaria Elimination Programme of the Government of Nigeria (NMEP) and financial support from the BMGF. The primary purpose of the study is to provide evidence of the impact of PMC on malaria burden and related clinical outcomes, and its operational feasibility for policy decision and the inclusion of PMC into upcoming programme and funding cycles for its National Malaria Control Strategic Plan. The objectives are:

1. To evaluate the impact of PMC in children aged 2-18 months on key child health outcomes including malaria burden, hospitalisations, and anaemia.
2. To describe indicators of operational feasibility of PMC by identification and measurement of key determinants of successful uptake and implementation of PMC.

DETAILED DESCRIPTION:
Study Design and Procedures The impact of PMC will be evaluated in a two-arm cluster-randomised controlled trial and nested case control study. The primary impact outcomes are a comparison of the incidence of clinical malaria in children 2-18 months of age visiting selected sentinel primary care facilities in intervention arm and comparison (standard care) arm wards in the study site, and the protective effectiveness of SP in the 28 days following a dose in intervention arm wards. A ward, the lowest level of health services administration for the State, will be the cluster unit of randomisation. A single facility meeting study eligibility criteria will be selected in each ward as the sentinel facility in which study outcomes will be evaluated (bi-monthly extraction of data on confirmed malaria cases by the study team). Strengthened age recording (full age in months) of visiting children will be implemented in each sentinel facility. An identical programme of data collection will take place in secondary and tertiary hospitals which serve the study site and will include data on admissions of children with an address in a study ward.

Cross sectional household 'malariometric' surveys will be conducted in catchment area communities of ;in both arms at baseline, at 18 months following start of PMC implementation, and at 24 months once implementation ends. Data on coverage of PMC doses (main indicator of feasibility) will be collected from child health record cards or caregiver report for children in the age groups eligible to receive the doses in question. Additional data on malaria infection (RDT test) and anaemia prevalence will be collected during the cross sectional surveys.

Collection of malaria data from sentinel facilities for children aged 19 months and older who were eligible to receive PMC during the implementation period (but too old at the end of implementation) will continue for an additional 12 months following the end of implementation period. The potential rebound effects of the intervention will be assessed in this period by a comparison of incidence rates in control and intervention arm wards.

Sample size (impact): The expected reduction in incidence of malaria in children aged 2-18 months after 18 months of implementation is conservatively estimated to be between 18%-32% contingent on the level of coverage of PMC doses in the intervention arm; enrolling 40 wards in each arm (for a total of 80) will provide 90% power to detect an impact of 20% in this age group after 18 months of implementation, and 95% after 24 months of implementation. We will also recruit children aged 2-18m with clinical malaria from 8 of the 40 intervention arm sentinel facilities and match these to 2-4 controls to have 95% power to detect a protective effectiveness of 50% reduction in malaria in the 28 days following a dose of SP.

Sample size (feasibility): To estimate coverage for any dose of 50% with a margin of error of 8%, assuming a design effect of 2.44 based on an implied intra cluster correlation coefficient of 0.18 (Nigeria DHS) to account for the cluster sample strategy, and allowing for 10% non-response, 25 children aged 2-36 months will be required in each cluster (ward), for a total of 25x40=1,000 in each arm of the study and with a total of 2000 across both arms.

Follow-up period: The total follow-up period of implementation will be 24 months, starting April 2023 to March 2025. The primary evaluation of impact and feasibility will occur in the first 18 months of implementation (April 2023 - September 2024).

Description of intervention: Health facility staff will be trained to offer scheduled doses of SP linked to the EPI delivery platform in children aged 10 weeks to 15 months (six doses), plus additional 'pragmatic' monthly doses offered outside of the EPI schedule to children up to 18 months of age (up to eleven additional doses). Additional social mobilisation and social behaviour change (SBC) activities will be conducted throughout the implementation period to increase demand and uptake of vaccination and PMC services in the study population.

Pharmacovigilance: Spontaneous (passive) adverse event (AE) reporting will be implemented in all study facilities (both sentinel and non-sentinel facilities in study wards),and will include training of health facility staff to recognise and manage known potential side effects of SP, and the development of picture based AE cards and posters for families and facility staff. Children with severe AEs will be referred to secondary/tertiary facilities as appropriate. A programme of active AE monitoring in a cohort of children will be additionally implemented in 2 facilities in each intervention arm in order to collect more detailed data on timings and symptoms following PMC or EPI doses, and to compare AE reporting rates between arms.

Additional activities: Cross-sectional health facility surveys and stakeholder interviews will take place during the follow-up period to collect data on implementation outcomes, alongside qualitative data collection in focus group discussions and in-depth interviews.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 weeks to 24 months
* Healthy

Exclusion Criteria:

* severe acute malnutrition, or
* allergic to sulphur containing medication,
* HIV positive,
* taking cotrimoxazole as prophylaxis or treatment, or SP, or other sulphur-containing medication in the previous 4 weeks, and
* children with a positive malaria RDT

Ages: 10 Weeks to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-08-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
. Incidence rate of clinical malaria | 18 months
  Incidence rate of parasitologically-confirmed clinical malaria cases in children 2-18 months presenting to selected sentinel facilities over 18 months* of implementation.
Protective effectiveness of SP | 18 months
  Protective effectiveness of SP treatments as measured by the percentage reduction in the incidence of malaria associated with receipt of SP in the last 28 days over 18 months* of implementation

SECONDARY OUTCOMES:
Prevalence of malaria infection | 18 months
  Prevalence of reported malaria in eligible children aged 2-18 months visited in an endline cross-sectional survey after 18m of implementation.
Prevalence of anaemia | 18 months
  Prevalence of anaemia (haemoglobin <80g/L) in eligible children aged 2-18 months visited in an endline cross-sectional survey after 18m of implementation.
Incidence rate of all-cause hospitalisations | 18 months
  Incidence of all-cause hospitalisations in eligible children aged 2-18 months with an address in a study ward, collected from hospital registration records over 18 months* of implementation.
Incidence rate of clinical malaria (rebound period) | 12 months following implementation
  Incidence rate of parasitologically-confirmed clinical malaria cases in children aged 19-36 months presenting to selected sentinel facilities in the 12 months following the end of the implementation period
Coverage of scheduled SP doses | 18 months
  For each of six scheduled doses of SP, the percentage of children who received the dose in question on time or within 4 weeks following the scheduled date will be estimated for children meeting age-eligibility criteria for each dose, in a cross sectional survey after 18 months* of implementation
Coverage of vaccine or vitamin A doses | 18 months of implementation
  For each EPI timepoint, the percentage of children who received the vaccine/supplement in question in will be estimated for children meeting age-eligibility criteria for each dose, in a cross sectional survey after 18 months* of implementation
Acceptability of PMC | 18 month
  Mean PMC acceptability score using an appropriate validated instrument (Acceptability of Intervention Measure - AIM), given by caregivers of eligible children in the intervention arm, measured during the endline cross-sectional survey after 18m of implementation. (intervention arms only) Mean PMC acceptability score using an appropriate validated instrument (Acceptability of Intervention Measure - AIM[Weiner et al 2017]" The instrument is validated in short form to gauge respondent acceptance of a programme by answering 4 direct questions. Minimum and maximum values for this measure are 4 and 20.
Integration of PMC into EPI delivery platform | 18 months
  Percentage of children visited in an endline cross-sectional survey who were eligible to receive SP and vaccines or vitamin A at a scheduled visit who received both an SP dose and the appropriate vaccine or Vitamin A on the same day. (intervention arms only)
Appropriateness of PMC | 18 months
  Mean appropriateness of PMC score using a suitable validated instrument (Intervention Appropriateness Measure - IAM27), given by policymakers at local (facility), state and national level interviewed at the end of follow-up. Mean appropriateness of PMC score using a suitable validated instrument (Intervention Appropriateness Measure - IAM[Weiner et al 2017]").
  The instrument is validated in short form to gauge degree of appropriateness (perspective of respondent) of a programme by answering 4 direct questions. Minimum and maximum values for this measure are 4 and 20.
  No cut-off scores for these instruments have been validated so it is recommended that full or mean scores are compared.
Fidelity of PMC delivery | 18months
  Mean health worker performance score based on a checklist-based survey of in-person observations of facility staff delivering PMC. (intervention arm only) Mean health worker performance score based on a checklist-based survey of in-person observations of facility[/and CHW] staff delivering PMC" using WHO health facility Survey manual.
  Min=0 max=100
. Adoption of PMC by facilities | 18 months
  Percentage of eligible intervention arm facilities surveyed that provided PMC services to children in the last 28 days. (intervention arms only)

CONTACTS AND LOCATIONS:
Overall Officials: James Tibenderana, PhD, Principal Investigator — Malaria Consortium
Locations (1):
- Ministry of Health, Oshogbo, Osun State, Nigeria